CLINICAL TRIAL: NCT00728195
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of 3 Fixed Doses of JNJ-37822681 Administered Twice Daily in Subjects With Schizophrenia
Brief Title: An Efficacy and Safety Study of 3 Fixed Doses of JNJ-37822681 in Participants With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014737; 37822681SCH2002; 2007-007083-22
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Central Nervous System; JNJ-37822681
MeSH Terms: conditions — Schizophrenia | interventions — N-(1-(3,4-difluorobenzyl)piperidin-4-yl)-6-(trifluoromethyl)pyridazin-3-amine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo First, Then Olanzapine (Placebo Comparator): Participants will receive 2 matching placebo capsules orally twice daily for 6 consecutive weeks, then 2 matching placebo capsules orally in the morning and olanzapine 10 milligram (mg) capsule along with matching placebo capsule orally in the evening for next 1 week, then 2 matching placebo capsules orally in the morning and olanzapine 10 mg capsule along with olanzapine 5 mg capsule orally in the evening for next 5 weeks.
  Interventions: Drug: Olanzapine; Drug: Placebo
- JNJ-37822681 10 mg (Experimental): Participants will receive 1 matching placebo capsule along with JNJ-37822681 10 mg capsule orally twice a day for 12 consecutive weeks.
  Interventions: Drug: JNJ-37822681; Drug: Placebo
- JNJ-37822681 20 mg (Experimental): Participants will receive 1 matching placebo capsule along with JNJ-37822681 20 mg capsule orally twice a day for 12 consecutive weeks.
  Interventions: Drug: JNJ-37822681; Drug: Placebo
- JNJ-37822681 30 mg (Experimental): Participants will receive JNJ-37822681 30 mg (one 10 mg capsule along with JNJ-37822681 20 mg capsule) orally twice a day for 12 consecutive weeks.
  Interventions: Drug: JNJ-37822681
- Olanzapine (Active Comparator): Participants will receive 2 matching placebo capsules orally in the morning and olanzapine 10 mg capsule along with matching placebo capsule orally in the evening for 1 week, then 2 matching placebo capsules orally in the morning and olanzapine 10 mg capsule along with olanzapine 5 mg capsule orally in the evening for next 11 consecutive weeks.
  Interventions: Drug: Olanzapine; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-37822681 — Participants will receive JNJ-37822681 capsule 10 mg orally twice a day for 12 consecutive weeks.
  Arms: JNJ-37822681 10 mg
Drug: JNJ-37822681 — Participants will receive JNJ-37822681 capsule 20 mg orally twice a day for 12 consecutive weeks.
  Arms: JNJ-37822681 20 mg
Drug: JNJ-37822681 — Participants will receive JNJ-37822681 capsule 30 mg orally twice a day for 12 consecutive weeks.
  Arms: JNJ-37822681 30 mg
Drug: Olanzapine — Participants will receive olanzapine 10 mg capsule alone or in combination with olanzapine 5 mg capsule orally for 6 or 12 weeks.
  Arms: Olanzapine; Placebo First, Then Olanzapine
Drug: Placebo — Participants will receive matching placebo capsules orally for 12 weeks.
  Arms: JNJ-37822681 10 mg; JNJ-37822681 20 mg; Olanzapine; Placebo First, Then Olanzapine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 3 fixed doses of JNJ-37822681 compared with placebo (an inactive substance that is compared with a drug to test if the drug has a real effect in a clinical trial) after 6 weeks treatment and olanzapine after 12 weeks treatment in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), double-blind (neither the participant nor the physician know the study medication drug name), randomized (study drug assigned by chance), placebo- and active-controlled, parallel-group (a clinical trial comparing the response in two or more groups of participants receiving different treatments), dose-response study in participants with schizophrenia. The total study duration will not exceed 16 weeks for each participant and will include following visits: screening, baseline, Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 11 and 13 (end of treatment or early withdrawal), and a post-study safety visit (1 week after final dose of study drug). All participants will be hospitalized during the first 2 weeks of treatment for detailed follow-up of safety and disease status. Following a screening period, participants will be randomly assigned to one of 5 treatment groups to receive oral doses of JNJ-37822681 (10, 20 or 30 milligram [mg] twice a day) for 12 weeks, olanzapine 15 mg daily for 12 weeks, or placebo for 6 weeks followed by olanzapine 15 mg daily for the remaining 6 weeks. Olanzapine will be initiated at 10 mg daily for 1 week and then increased to 15 mg daily for the remainder of the treatment period. Efficacy will primarily be evaluated by Positive And Negative Syndrome Scale (PANSS). Participants' safety will also be monitored at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been diagnosed with schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) (295.10, 295.20, 295.30, 295.60, 295.90) at least 1 year prior to screening
* Participants must be experiencing an acute (a quick and severe form of illness in its early stage) exacerbation of less than 6 months duration, with a Positive and Negative Syndrome Scale (PANSS) total score at screening between 70 and 120 inclusive and at baseline of between 60 and 120 inclusive
* Women of child bearing potential must have a negative urine pregnancy test at screening and baseline before receiving the study drug
* Participants must agree to voluntary hospitalization for a minimum of 14 days
* BMI (Body Mass Index) maximum 40 kilogram per meter square (kg/m^2), inclusive (BMI=weight/height^2)

Exclusion Criteria:

* A DSM-IV axis I diagnosis other than schizophrenia
* A DSM-IV diagnosis of substance dependence within 6 months prior to screening evaluation
* Any clinically relevant medical condition that could potentially alter the absorption (the way a drug or other substance enters the body), metabolism, or excretion (the way that substances leave the body) of the study medication, such as Crohn's disease (serious inflammation of any part of the gastrointestinal tract), liver disease, or renal (pertaining to the kidneys) disease
* Relevant history of any significant and/or unstable cardiovascular (pertaining to the heart and blood vessels), respiratory, neurological (including seizures) or significant cerebrovascular (pertaining to brain and blood vessels), renal, hepatic, endocrine (pertaining to the glands that make hormones), or immunologic diseases
* History of neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6 | Baseline and Week 6
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). The total score ranges from 30 to 210 and higher score indicates greater severity.

SECONDARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Subscale Scores at Week 6 and 12 | Baseline, Week 6 and 12
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The PANSS provides a total score and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each item scored on a scale of 1 (absent) to 7 (extreme). Positive subscale score ranges from 7 (absent) to 49 (extreme psychopathology), negative subscale score ranges from 7 (absent) to 49 (extreme psychopathology) and general psychopathology subscale score ranges from 16 (absent) to 112 (extreme psychopathology).
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Subscale Scores at Week 6 and 12 | Baseline, Week 6 and 12
  The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consists of 7 items with total score range of 7-49 and uncontrolled hostility/excitement (UHE) subscale and anxiety/depression subscale, each consists of 4 items with total score range of 4-28. Higher score indicates greater severity.
Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 6 and 12 | Baseline, Week 6 and 12
  The CGI-S rating scale assesses the severity of a participant's overall clinical condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe).
Change From Baseline in Subjective Well-Being on Neuroleptics (SWN) Total Score at Week 6 and 12 | Baseline, Week 6 and 12
  The SWN is a participant self rated scale to evaluate the participant's feelings during the past 7 days on a form with 20 statements, subsequently divided into 5 subscales: mental-functioning, self-control, emotional regulation, physical functioning and social integration. Each item is scored between 1 (not at all) and 6 (very much). Total score ranges from 20-120 with higher scores indicating higher subjective well-being.
Change From Baseline in Nurses' Observation Scale for Inpatient Evaluation (NOSIE) Total Score at Week 2 | Baseline and Week 2
  The NOSIE comprises 30 items which form 6 scales: social competence, social interest, personal neatness, irritability, manifest psychosis and retardation and is completed by a suitably trained and experienced member of the nursing staff. Each item is scored from 0 (never) to 4 (always). It was assessed only at 2 weeks when the participants were hospitalized. Total score ranges from 0 to 120, with lower score indicating better results.
Change From Baseline in Plasma Markers Level for Lipid and Glucose Metabolism at Week 6 and 12 | Baseline, Week 6 and 12
  Change from baseline in the level of plasma (liquid part of blood where cells float) markers for lipid (fat) and glucose (type of sugar found in the blood) metabolism (process of breaking down substances in the cells to obtain energy) is calculated. Markers for lipid metabolism include fasting total cholesterol, high-density lipoproteins (HDL), low-density lipoproteins (LDL), very low-density lipoproteins (VLDL), triglycerides and free fatty acids. Fasting glucose level is used as marker for glucose metabolism.
Change From Baseline in Free Fatty Acids Level at Week 6 and 12 | Baseline, Week 6 and 12
  Change from baseline in the level of free fatty acids (plasma marker for lipid metabolism) is calculated.
Change From Baseline in Insulin Level at Week 6 and 12 | Baseline, Week 6 and 12
  Change from baseline in the level of insulin (the hormone that controls blood sugar levels) as plasma marker for glucose metabolism is calculated.
Change From Baseline in Glycosylated Hemoglobin (HbA1c) Level at Week 6 and 12 | Baseline, Week 6 and 12
  Change from baseline in the level of glycosylated hemoglobin (substance that carries oxygen and gives blood its red color) as plasma marker for glucose metabolism is calculated.
Change From Baseline in Body Mass Index (BMI) at Week 6 and 12 | Baseline, Week 6 and 12
  The BMI is calculated by dividing the weight (in kilogram) by square of height (in meters).
Change From Baseline in Body Weight at Week 6 and 12 | Baseline, Week 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (45):
- Bulgaria (5):
  - Burgas
  - Pazardzhik
  - Radnevo
  - Rousse
  - Sofia
- Estonia (2):
  - Tallinn
  - Tartu
- Lithuania (2):
  - Kaunas
  - Vilnius
- Malaysia (3):
  - Johor Bahru
  - Kuala Lumpur
  - Kuching
- Romania (7):
  - Arad
  - Brasov
  - Bucharest
  - Jebel
  - Oradea
  - Sibiu
  - Tg Mures
- Russia (9):
  - Ekaterinburg Na
  - Moscow
  - Moscow Russia
  - N Novgorod Na
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk Na
  - Yaroslavl
- South Africa (3):
  - Cape Town
  - Centurion Gauteng
  - Pretoria
- South Korea (4):
  - Gwangju
  - Gyeongsangnam-Do
  - Incheon
  - Seoul
- Taiwan (3):
  - Hualien City
  - Kaohsiung City
  - Taipei
- Ukraine (7):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kherson
  - Kiev
  - Odesa
  - Simferopol

REFERENCES:
- [Derived] Anghelescu IG, Janssens L, Kent J, de Boer P, Tritsmans L, Daly EJ, van Nueten L, Schmidt ME. Does early improvement predict response to the fast-dissociating D(2) receptor antagonist JNJ-37822681 in patients with acute schizophrenia? Eur Neuropsychopharmacol. 2013 Sep;23(9):1043-50. doi: 10.1016/j.euroneuro.2012.08.017. Epub 2012 Sep 18. PMID 22995972
- See also: A Randomized, Double Blind, Placebo and Active Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of 3 Fixed Doses of JNJ 37822681 Administered Twice Daily in Subjects with Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=778&filename=CR014737_CSR.pdf